CLINICAL TRIAL: NCT07018050
Title: A Multicenter, Open-Label Phase II Study to Evaluate QLS32015 Combination Therapy in the Treatment of Multiple Myeloma
Brief Title: Phase II Study of QLS32015 Combination Therapy in the Treatment of Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLS32015-202
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-05

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — pomalidomide; Dexamethasone; daratumumab; Bortezomib; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QLS32015(SC) in combination with Pomalidomide (Experimental): Participants will receive QLS32015 as SC injections; Pomalidomide will be self-administered as a single dose orally; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug.
  Interventions: Drug: QLS32015; Drug: Pomalidomide; Drug: Dexamethasone
- QLS32015(SC) in combination with QL2109 or Daratumumab. (Experimental): Participants will receive QLS32015 and QL2109 or Daratumumab as SC injections; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug.
  Interventions: Drug: QLS32015; Drug: Dexamethasone; Drug: QL2109 or Daratumumab
- QLS32015(SC) in combination with QL2109 or Daratumumab and Pomalidomide (Experimental): Participants will receive QLS32015 and QL2109 or Daratumumab as SC injections; Pomalidomide will be self-administered as a single dose orally; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug
  Interventions: Drug: QLS32015; Drug: Pomalidomide; Drug: Dexamethasone; Drug: QL2109 or Daratumumab
- QLS32015(SC) in combination with Bortezomib for injection and Lenalidomide (Experimental): Participants will receive QLS32015 and Bortezomib as SC injections; Lenalidomide will be self-administered as a single dose orally; dexamethasone may be given orally or intravenously as a pretreatment medication and study drug
  Interventions: Drug: QLS32015; Drug: Dexamethasone; Drug: Bortezomib; Drug: Lenalidomide

INTERVENTIONS:
Drug: QLS32015 — QLS32015 will be administered subcutaneously
Drug: Pomalidomide — Pomalidomide will be self-administered as a single dose orally
  Arms: QLS32015(SC) in combination with Pomalidomide; QLS32015(SC) in combination with QL2109 or Daratumumab and Pomalidomide
Drug: Dexamethasone — Dexamethasone will be administered orally or intravenously
Drug: QL2109 or Daratumumab — QL2109 or Daratumumab will be administered subcutaneously.
  Arms: QLS32015(SC) in combination with QL2109 or Daratumumab and Pomalidomide; QLS32015(SC) in combination with QL2109 or Daratumumab.
Drug: Bortezomib — Bortezomib will be administered subcutaneously
  Arms: QLS32015(SC) in combination with Bortezomib for injection and Lenalidomide
Drug: Lenalidomide — Lenalidomide will be self-administered as a single dose orally
  Arms: QLS32015(SC) in combination with Bortezomib for injection and Lenalidomide

SUMMARY:
The purpose of the study is to compare the efficacy of QLS32105 (SC) in combination with Pomalidomide, and QLS32105 (SC) in combination with QL2109 or Daratumumab, and QLS32105 (SC) in combination with QL2109 or Daratumumab and Pomalidomide, and QLS32105(SC) in combination with Bortezomib and Lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma confirmed according to the 2016 International Myeloma Working Group (IMWG) diagnostic criteria;
* Prior therapy: Relapsed, progressed, or intolerant to ≥1 prior line of anti-multiple myeloma therapy;
* Measurable disease at screening, defined by at least one of the following:

  * Serum M-protein ≥1.0 g/dL (10 g/L);
  * Urine M-protein ≥200 mg/24 hours;
  * Serum immunoglobulin free light chain ≥10 mg/dL (100 mg/L) with an abnormal serum immunoglobulin κ/λ free light chain ratio.

Exclusion Criteria:

* History of Grade 3 or higher cytokine release syndrome (CRS) associated with any T-cell redirecting therapy (e.g., CD3-redirecting technologies or CAR-T cell therapy);
* Prior anti-myeloma therapies within the specified timeframes before enrollment:

  * Previous treatment with GPRC5D-targeted therapy;
  * Genetically modified adoptive cell therapy (e.g., chimeric antigen receptor T-cell [CAR-T], natural killer [NK] cell therapy) within 3 months;
  * Targeted therapy, investigational drugs, or invasive investigational medical devices within 21 days or 5 half-lives (whichever is longer);
  * Monoclonal antibodies or bispecific antibody therapy for multiple myeloma within 21 days or 5 half-lives (whichever is longer);
  * Cytotoxic therapy within 21 days;
  * Proteasome inhibitor therapy within 14 days;
  * Immunomodulatory drug therapy within 7 days;
* Radiotherapy within 14 days (except low-dose palliative radiation [10-30 Gy]);
* Prior intolerance to Pomalidomide (applies to treatment cohorts containing Pomalidomide);
* Prior intolerance to Bortezomib (applies to treatment cohorts containing bortezomid);
* Prior intolerance to Lenalidomide (applies to treatment cohorts containing Lenalidomide);
* Prior intolerance to Daratumumab (applies to treatment cohorts containing Daratumumab).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
ORR (Partial Response [PR] or Better) | Up to 2 years
  Overall response (PR or better) is defined as percentage of participants who have a PR or better per International Myeloma Working Group (IMWG) criteria
Overall Minimal Residual Disease (MRD) | Up to 2 years
  MRD-negative is defined as proportion of participants who achieve MRD negativity at a threshold of 10^-5 at any timepoint after the first dose of study drug and before disease progression or start of subsequent antimyeloma therapy

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as time from the date of randomization to the first documentation of disease progression, or death due to any cause, whichever is reported first

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China